CLINICAL TRIAL: NCT06027398
Title: Efficacy of SARS-COV-2 Detection From Used Surgical Mask Compared to Standard Detection Method
Brief Title: SARS-COV-2 Detection From Used Surgical Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 138/64
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2 Virus
Keywords: Nasopharyngeal swab; RT-PCR; SARS-CoV-2; surgical mask

STUDY DESIGN:
Intervention Model Description: To compare the efficacy of SARS-CoV-2 RNA detection from used surgical masks with standard detection methods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-CoV-2 RNA in masks (Experimental): . After the participants had worn the masks for 8 h, the nurse collected the filters and placed each into a viral transport medium (VTM) tube This was placed inside a clean plastic bag, sprayed with alcohol, placed in an icebox and sent to the biomolecular laboratory for real-time RT-PCR SARS-CoV-2 testing.
  Interventions: Diagnostic Test: SARS-CoV-2 RNA detection

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 RNA detection — SARS-CoV-2 RNA detection in used mask filters

SUMMARY:
The real-time reverse transcription-polymerase chain reaction (RT-PCR) test is regarded as the gold standard for SARS-CoV-2 detection. Proper specimen collection and obtaining a sufficient sample are the most important steps for laboratory diagnosis. The nasopharyngeal (NP) swab is recommended as the reference collection method. However, NP swab collection is invasive and uncomfortable for patients and poses some risk to healthcare workers. This study aimed to compare the efficacy of SARS-CoV-2 RNA detection from used surgical masks with the NP swab method using RT-PCR testing

DETAILED DESCRIPTION:
Proper specimen collection and obtaining sufficient samples are the most important steps for laboratory diagnosis of an infectious disease. Improper collection may lead to false or inconclusive test results. During the early stages of the COVID-19 outbreak, the Center for Disease Prevention and Control recommended collecting and testing an upper respiratory specimen [4]. Nasopharyngeal (NP) and oropharyngeal (OP) swabs are the preferred choice for initial SARS-CoV-2 diagnostic testing.

This study aimed to compare the efficacy of SARS-CoV-2 RNA detection from used surgical masks with standard detection methods. We tested for SARS-CoV-2 RNA in masks from patients with COVID-19 that had been worn for eight hours and compared this with NP swabs using RT-PCR testing. Hospitalized patients with laboratory-confirmed COVID-19 were recruited to provide surgical masks. Collection of used surgical mask samples by patients themselves is easy, convenient, requires no sampling equipment and decreases the risk of healthcare personnel exposure to COVID-19. If SARS-CoV-2 RNA can be detected on used surgical mask samples, this may encourage patients to provide specimens for testing and help in early detection and transmission prevention. As an alternative method to NP swabs, it may facilitate timely diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly confirmed SARS-CoV-2 positive cases admitted to a field hospital within 48 hours or outpatient with a positive result for SARS-CoV-2
* Should be able to wear a mask for 8 h according to the protocol

Exclusion Criteria:

* require oxygen intubation or any breathing support devices

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 269 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
the efficacy of SARS-CoV-2 RNA detection from used surgical masks | 3 months
  tested for SARS-CoV-2 RNA in masks from patients with COVID-19 that had been worn for eight hours and compared this with NP swabs using RT-PCR testing

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Principal Investigator — Navamindradhiraj University
Locations (1):
- 2 Division of Nephrology,Department of Medicine Pramongkutklao Hospital and College of Medicine,Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The data underlying this article are available in figshare 10.6084/m9.figshare.24064218
Supporting Information: SAP

REFERENCES:
- [Result] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Result] Gao Q, Bao L, Mao H, Wang L, Xu K, Yang M, Li Y, Zhu L, Wang N, Lv Z, Gao H, Ge X, Kan B, Hu Y, Liu J, Cai F, Jiang D, Yin Y, Qin C, Li J, Gong X, Lou X, Shi W, Wu D, Zhang H, Zhu L, Deng W, Li Y, Lu J, Li C, Wang X, Yin W, Zhang Y, Qin C. Development of an inactivated vaccine candidate for SARS-CoV-2. Science. 2020 Jul 3;369(6499):77-81. doi: 10.1126/science.abc1932. Epub 2020 May 6. PMID 32376603
- [Result] Qian Y, Zeng T, Wang H, Xu M, Chen J, Hu N, Chen D, Liu Y. Safety management of nasopharyngeal specimen collection from suspected cases of coronavirus disease 2019. Int J Nurs Sci. 2020 Apr 4;7(2):153-156. doi: 10.1016/j.ijnss.2020.03.012. eCollection 2020 Apr 10. PMID 32292635
- [Result] Comber L, Walsh KA, Jordan K, O'Brien KK, Clyne B, Teljeur C, Drummond L, Carty PG, De Gascun CF, Smith SM, Harrington P, Ryan M, O'Neill M. Alternative clinical specimens for the detection of SARS-CoV-2: A rapid review. Rev Med Virol. 2021 Jul;31(4):e2185. doi: 10.1002/rmv.2185. Epub 2020 Oct 22. PMID 33091200